CLINICAL TRIAL: NCT01419041
Title: A Phase I, Single Dose, Parallel-Group Study To Evaluate The Pharmacokinetics Of Crizotinib (PF-02341066) In Subjects With Impaired Renal Function
Brief Title: A Study to Evaluate The Pharmacokinetics Of Crizotinib (PF-02341066) In Subjects With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A8081020
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Renal Impairment
Keywords: renal impairment; crizotinib; pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Other): CLCR: Creatinine clearance
  Interventions: Drug: crizotinib
- Arm B (Other): CLCR: Creatinine clearance
  Interventions: Drug: crizotinib

INTERVENTIONS:
Drug: crizotinib — Single-dose oral 250 mg crizotinib in subjects with normal renal function (CLcr =>90 mL/min)
  Arms: Arm A
Drug: crizotinib — Single-dose oral 250 mg crizotinib in subjects with severe renal impairment (CLcr <30 mL/min)
  Arms: Arm B

SUMMARY:
The present study is being conducted to evaluate whether or not severe renal impairment has an effect on crizotinib Pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

All Subjects

* Healthy male and/or female of non childbearing potential subjects between the ages of 18 and 65 years, inclusive ('healthy' is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG, and clinical laboratory tests).
* Body Mass Index (BMI) of 18 to 40 kg/m2 inclusive; and a total body weight >50 kg (>110 lbs).

Subjects with Normal Renal Function (Group 1)

* Normal renal function (CLcr =>90 mL/min) during the screening period.
* Matched 1-to-1 to subjects in Group 2 with respect to age (+/-5 years), weight (+/-10 kg), gender, and race according to protocol.

Subjects with Severe Renal Impairment (Groups 2)

* Good general health commensurate with the population with chronic kidney disease.
* Severe renal impairment (CLcr<30 mL/min) during the screening period.

Exclusion Criteria:

All Subjects

* Renal allograft recipients.
* Any condition possibly affecting drug absorption.
* 12 lead ECG demonstrating QTc >470 msec at screening.
* Urinary incontinence without catheterization.
* A positive urine drug screen.
* History of regular alcohol consumption.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half lives preceding the first dose of study medication.
* Pregnant or nursing females; females of childbearing potential, including those with tubal ligation.
* Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing.

Subjects with Severe Renal Impairment (Groups 2)

* Subjects with any significant hepatic, cardiac or pulmonary disease (apart from stable ischemic heart disease), or subjects who are clinically nephrotic.
* Subjects requiring hemodialysis.
* Subjects with strict fluid restriction (ie, <1500 mL/24 hours).
* Significant bleeding diathesis which could preclude multiple venipuncture.
* Use of food or drugs that are CYP3A4 inhibitors and inducers.
* Herbal supplements and hormone replacement therapy must be discontinued 28 days prior to the first dose of trial medication
* Concurrent use of drugs that are CYP3A4 substrates with narrow therapeutic indices.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Plasma AUCinf (Area under the plasma concentration versus time curve from zero to infinity) for crizotinib | 18 months
Plasma Cmax (Maximum plasma concentration) for crizotinib | 18 months

SECONDARY OUTCOMES:
Plasma AUClast (Area under the plasma concentration versus time curve from zero to the last quantifiable concentration) for crizotinib | 18 months
Tmax (Time to Cmax) for crizotinib | 18 months
t1/2 (terminal half-life) for crizotinib | 18 months
CL/F (Apparent oral clearance) for crizotinib | 18 months
Vz/F (Apparent volume of distribution after oral dose) for crizotinib | 18 months
fu (fraction of unbound drug in plasma) for crizotinib | 18 months
AUCinf,u (unbound AUCinf) for crizotinib | 18 months
AUClast,u (unbound AUClast) for crizotinib | 18 months
Cmax,u (unbound Cmax) for crizotinib | 18 months
CL/Fu (unbound apparent oral clearance) for crizotinib | 18 months
CLR (Renal clearance) for crizotinib | 18 months
Ae (Cumulative amount of drug recovered unchanged in the urine) for crizotinib | 18 months
Ae% (Cumulative amount of drug recovered unchanged in the urine expressed as fraction of administered dose) for crizotinib | 18 months
AUCinf (Area under the plasma concentration versus time curve from zero to infinity) for PF-06260182 | 18 months
AUClast (Area under the plasma concentration versus time curve from zero to the last quantifiable concentration) for PF-06260182 | 18 months
Cmax (Maximum plasma concentration) for PF-06260182 | 18 months
Tmax (Time to Cmax) for PF-06260182 | 18 months
t1/2 (terminal half-life) for PF-06260182 | 18 months
fu (fraction of unbound drug in plasma) for PF-06260182 | 18 months
AUCinf,u (unbound AUCinf) for PF-06260182 | 18 months
AUClast,u (unbound AUClast) for PF-06260182 | 18 months
Cmax,u (unbound Cmax) for PF-06260182 | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Saint Paul, Minnesota

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081020&StudyName=A%20Study%20to%20Evaluate%20The%20Pharmacokinetics%20Of%20Crizotinib%20%28PF-02341066%29%20In%20Subjects%20With%20Impaired%20Renal%20Function%20